CLINICAL TRIAL: NCT04660864
Title: Nasal Cavity Cooling for the Symptomatic Relief of Migraine Headache - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: BrainCool (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-05471
Record Dates: First submitted 2020-11-17; First posted 2020-12-09 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Single group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rhinochill (Experimental): Treatment with nasal cavity cooling 10 minutes during three consecutive migraine attacks.
  Interventions: Device: Nasal cavity cooling device.

INTERVENTIONS:
Device: Nasal cavity cooling device. — The RhinoChill® system cools by intranasal evaporation of a liquid coolant sprayed onto the surface of the nasal cavity. The RhinoChill® system is intended for use for the relief of pain and symptoms associated with acute migraine attack.

SUMMARY:
The aim of the study is to evaluate the effect of self-administered intranasal cooling for the symptomatic relief of migraine headache and associated symptoms in an "at home setting".

10-20 patients - who have been diagnosed according to the International Classification of Headache disorders (2nd Edition) criteria for Episodic migraine, with or without aura - will be included in the study.

During a screening period of one month participants will record their migraine symptoms, any treatment and treatment effects. After a minimum om two migraine attacks the participants receive individual instructions on how to use the The RhinoChill® system. During the following treatment period of the study, participants are instructed to treat their upcoming three migraine attacks with 10 minutes of nasal cavity cooling according to the instructions and thereby register symptoms and treatment effects after 10 minutes, 1 hour, 2 hours, 24 hours and 48 hours.

DETAILED DESCRIPTION:
Mechanical techniques to alleviate migraine symptoms have been used for many years, cooling and compression being the most frequently applied. Cryotherapy is the most common non-pharmacological self-administered pain-relieving method currently used by migraine sufferers.

The RhinoChill® System is a CE-Marked device that is currently commercially available in Europe. The RhinoChill® device is intended for temperature reduction in patients via the nasal cavity and can be used across a range of medical and surgical indications where reduction in patient temperature is required. The RhinoChill® system was originally designed specifically for use in the pre-hospital, in-hospital, in-clinic or other clinical settings for the induction of therapeutic hypothermia (reduction in brain and body temperature to between 32-34oC), in which other commercial cooling systems are not practical for use. The RhinoChill® system is portable and runs on batteries. The system cools by spraying an evaporative coolant into the nasal cavity via intranasal catheters. A previous study has shown that the use of RhinoChill® intranasal cooling within a clinic environment provided a statistically significant reduction of pain and associated symptoms of migraine at 5 and 10 minutes (during treatment) and at 1 and 2 hours following treatment along with significant effect on pain and symptoms at 24 hours (all p values <0.001).

The aim of the study is to evaluate the effect of intranasal cooling for the symptomatic relief of migraine headache and associated symptoms when the treatment is self-administered by the patient at home.

The proposed study will be single group assignment with treatment self-administered by patients in their own home, with support and oversight from research support staff working under the direction of the investigators.

The study process is as summarized:

Participants will be identified through adverts at Lund University and are able to register interest via telephone or email. They are then contacted by a researcher by telephone for a brief eligibility check and to book a first meeting at the Braincool office.

Meeting 1, at Braincool office (researcher and research support team):

* Eligibility check - stage one (Case Report Form 1)
* Trial information, viewing of device and catheter
* Informed Consent Form complete
* Instruction on how to register migraine attack symptoms and treatment effects in application/CRF2.

Screening period starts. When the participant has registered two migraine attacks during the screeing period the next meeting is booked:

Meeting 2, home visit (research support team):

o Training on how to use the RhinoChill® device safely and how to register migraine symptoms and treatment effects in application/CRF 3

During the following treatment period of the study, participants are instructed to treat their upcoming three migraine attacks with 10 minutes of nasal cavity cooling according to the instructions and thereby register symptoms and treatment effects after 10 minutes, 1 hour, 2 hours, 24 hours and 48 hours.

When the participant has used the RhinoChill® device to treat three episodes of migraine, or a duration of 3 months post-study has passed, the final meeting is booked.

Meeting 3, home visit (research support team):

* Collection of device and other equipment
* Evaluation on any side effects/adverse events/CRF 4.

ELIGIBILITY:
Inclusion Criteria:

* Meets the International Classification of Headache Disorders (2nd edition) criteria for episodic migraine, with or without aura.
* Migraine diagnosis >1 year
* Migraine attacks 2-8 times/month
* Living in Malmö-Lund area
* Reliable contraception (fertile women)

Exclusion Criteria:

* Any change of migraine prophylaxis within three months prior to study begin
* Failure of participant to adhere to protocol requirements
* Smoker or smoker in participants household
* Prior nose surgery or intranasal obstruction
* Pregnancy, breast feeding or planned pregnancy during trial period
* Oxygen dependency
* Medical history of skull base fracture or severe facial trauma
* No migraine attacks during prolonged screening phase (60 days)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Reduction of headache | 10 minutes after baseline (immediately after treatment) compared to baseline
  Scoring of headache on a 4-graded scale (none-mild-moderate-severe).
Reduction of nausea | 10 minutes after baseline (immediately after treatment) compared to baseline
  Scoring of symptoms on a 4-graded scale (none-mild-moderate-severe) regarding nausea
Reduction of photophobia | 10 minutes after baseline (immediately after treatment) compared to baseline
  Scoring of symptoms on a 4-graded scale (none-mild-moderate-severe) regarding photophobia
Reduction of phonophobia | 10 minutes after baseline (immediately after treatment) compared to baseline
  Scoring of symptoms on a 4-graded scale (none-mild-moderate-severe) regarding photophonia

SECONDARY OUTCOMES:
Headache response | Comparing baseline/before treatment and 1. immediately following treatment (10 minutes),2. 1 hour, 3. 2 hours and 4. 24 hours following treatment.
  The patient scores the headache symptoms on a 4-graded scale (none-mild-moderate-severe). Any improvement of pain is recorded.
Relapse incidence | Between 2-48 hours after intervention
  Frequency of headache returns
Sustained pain freedom, number of patients that sustain pain freedom 2-48 hours after intervention. | 2-48 hours after intervention
  pain free with no use of rescue medication or relapse
Impact on nausea | At baseline and 1, 2, 24 hours after treatment
  Scoring of symptoms none-mild-moderate-severe regarding nausea
Impact on photophobia | At baseline and 1, 2, 24 hours after treatment
  Scoring of symptoms none-mild-moderate-severe regarding photophobia
Impact on phonophobia | At baseline and 1, 2, 24 hours after treatment
  Scoring of symptoms none-mild-moderate-severe regarding , photophobia and phonophobia
Comparison of headache response between RhinoChill compared to standard treatment during screening period | Screening phase compared to intervention phase
  Comparison of average treatment effect on headache respons between standard treatment and intervention. Scoring of headache on a 10-graded scale, where higher values represents more pain
Average headache pain relief | At baseline and 10 minutes, 1, 2 and 24 hours after treatment.
  Scoring of pain on a 4-graded scale, (none-mild-moderate-severe) compared to baseline.
Tolerance to rhinochill cooling - pain | 10 minutes-1 hour
  Visual/analogue pain on a 10-graded scale, where higher values represents more pain.
Tolerance to rhinochill cooling - discomfort | 10 minutes-1 hour
  Visual/analogue discomfort score, on a 10-graded scale, where higher values represents more discomfort.
Adverse events | through study completion, an approximated average of 3 months.
  Any adverse events noted during the treatment, following treatment or during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Midlöv, Professor, Study Chair — Department of Clinical Sciences, Malmö, Lund University, Sweden; Moa Wolff, PhD, Principal Investigator — Department of Clinical Sciences, Malmö, Lund University, Sweden
Locations (1):
- Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanderpol J, Bishop B, Matharu M, Glencorse M. Therapeutic effect of intranasal evaporative cooling in patients with migraine: a pilot study. J Headache Pain. 2015 Jan 26;16:5. doi: 10.1186/1129-2377-16-5. PMID 25623151
- [Background] Ucler S, Coskun O, Inan LE, Kanatli Y. Cold Therapy in Migraine Patients: Open-label, Non-controlled, Pilot Study. Evid Based Complement Alternat Med. 2006 Dec;3(4):489-93. doi: 10.1093/ecam/nel035. Epub 2006 Jun 15. PMID 17173113